CLINICAL TRIAL: NCT04788602
Title: The Applications and Influences of Transthoracic Echocardiography in Stroke Patients
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202010048RINB
Record Dates: First submitted 2021-03-08; First posted 2021-03-09 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: the Impact of Echocardiography on the Recurrence of Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transthoracic echocardiography (TTE) is known to be an effective modality in assessing cardiac function as well as the structure of the heart. It was estimated that between 15% and 30% of ischemic strokes were due to a cardioembolic source, Therefore, TTE has been assumed as an important screening tool in patients with ischemic stroke, as atrial fibrillation is one of the leading risk factors. However, current guidelines have little evidence in whether performing TTE can alter clinical management and prevent a future stroke. We aim to present the association of performing TTE and clinical outcomes in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute stroke and receiving echocardiography

Exclusion Criteria:

* patients with acute stroke and not receiving echocardiography

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with acute stroke and receiving echocardiography
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
recurrent stroke | one year
  the correlation between the echocardiography and recurrence of stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency Medicine, National Taiwan University Hospital, Taipei, Taiwan